CLINICAL TRIAL: NCT05769270
Title: Development and Pilot RCT of a Telehealth-delivered Peer Navigation and Coping Skills Intervention to Increase PrEP Use in Young Black Men Who Have Sex With Men
Brief Title: Development of a Telehealth-delivered Peer Navigation and Coping Skills Intervention to Increase PrEP Use in Young Black MSM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator requested early termination of grant
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Fenway Community Health (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Calvin Fitch, PhD, Postdoctoral Fellow, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021P003220; 1K23MH129240 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-03-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hiv; Sexual Behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexual Behavior | interventions — Coping Skills; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Navigation and Coping Skills (Experimental): Participants will receive peer navigation and coping skills to increase PrEP use.
  Interventions: Behavioral: Peer Navigation and Coping Skills; Behavioral: Treatment as Usual
- Treatment as usual (Sham Comparator): Participants will receive referrals to PrEP and services.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Peer Navigation and Coping Skills — Participants will receive 6 sessions of peer navigation and coping skills
  Arms: Peer Navigation and Coping Skills
Behavioral: Treatment as Usual — Participants will receive referrals for PrEP and services

SUMMARY:
This proposal seeks to adapt an existing peer navigation protocol (by adding coping skills and using telehealth) to be feasible, acceptable, and capable of supporting both PrEP uptake and P-E adherence for YBMSM ages 15-24.

DETAILED DESCRIPTION:
Young Black men who have sex with men (YBMSM) ages 15-24 are heavily affected by HIV transmission and, at current rates, nearly half of Black MSM in the US will be infected with HIV in their lifetime. MSM represented 42% of all HIV diagnoses in Massachusetts from 2015-2017 and rates among Black MSM were 7 times that of White MSM. Fortunately, PrEP is highly effective at preventing HIV if adhered to in a prevention-effective (P-E) manner, which involves daily or event-based dosing specifically during periods of risk of HIV exposure (i.e., P-E adherence). Unfortunately, initiation and adherence among YBMSM is lower than other racial and age groups. According to Social Action Theory, barriers among YBMSM can be conceptualized as multifactorial, consisting of contextual factors (e.g., mood/arousal factors, structural factors, and demographics) and self-change processes (social interaction processes, motivations, generative capabilities, and problem-solving skills). An effective intervention must address contextual and self-change processes to promote PrEP uptake and P-E adherence.

The use of navigators (i.e., health workers trained to support ongoing adherence) has shown promise in promoting both PrEP uptake and sustained use in Black MSM by addressing structural barriers; however, rates of PrEP discontinuation were high. An NICHD-funded U01 study (SMILE) conducted in Boston found that peer navigation was highly acceptable for youth with HIV. The current study will use the Boston site of SMILE's peer navigation protocol. Notably, SMILE did not include behavioral components. In addition to structural barriers, YBSM often face unique barriers such as medical mistrust and disclosure concerns that affect self-change processes and impede PrEP uptake and P-E adherence. Limited knowledge exists on how these factors may impede PrEP use; however, it is clear these barriers may be addressed using problem/emotion-focused coping strategies. Many PrEP interventions require office visits, which may limit participation to those willing and able to present to a research office. Despite prevalent economic stressors, more than 90% of YMSM of color in various studies have smartphones, thus telehealth and remote study procedures may facilitate participation by YBMSM at highest HIV risk. This proposal seeks to adapt peer navigation from SMILE (adding coping skills and using telehealth) to be feasible, acceptable, and capable of supporting both PrEP uptake and P-E adherence for YBMSM ages 15-24.

Aim 1: Obtain qualitative knowledge on experiences of YBMSM ages 15-24 and specify role of peer navigator in promoting PrEP uptake and P-E adherence. I will conduct ~30 in-depth interviews with YBMSM at various stages of the PrEP continuum (e.g., never used, former user, and currently using PrEP) using a semi-structured interview guide. Interviews will explore how contextual factors and self-change processes influence PrEP uptake and P-E adherence. It will specify the role of a peer navigator (e.g., meeting frequency, demographics of navigator, topics to discuss and how best to employ technology-based tools and strategies). The knowledge gained from these interviews will be used to inform intervention development in Aim 2.

Aim 2: Develop and iteratively refine the intervention in consultation with a Youth Advisory Board Intervention development will be guided by Aim 1 findings and the IDEAS framework (i.e., generating ideas for intervention strategies, developing an initial intervention, gathering user feedback, and creating a viable intervention). We will recruit ~20 YBMSM via online and in-person strategies to participate in an advisory board meeting quarterly (virtually or in-person) to provide feedback on the intervention. The intervention will be iteratively refined after each meeting resulting in a refined intervention manual for use in the Aim 3 trial.

Aim 3: Evaluate the telehealth-delivered peer navigation/coping skills intervention for feasibility and acceptability. We will have a short, 3-month run-in of the intervention with 2-4 sexually active YBMSM, without HIV, ages 15-24. After further refinement, we will conduct a small (N=60) RCT of the peer navigation/coping skills intervention vs. treatment as usual (TAU; PrEP/case management referrals). The primary outcomes will be feasibility and acceptability. Secondarily, we will examine group differences in PrEP uptake, P-E adherence (proportion of covered sexual episodes), and sustained use at 6 months among those with risk. Outcomes of this aim will be a feasible (>75% enrollment; >75% of sessions attended) and acceptable (per questionnaires and exit interviews) intervention that can be tested in a larger efficacy trial in the context of a future R01 grant.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative (by self-report)
* Black race (of any ethnicity, by self-report)
* age 15-24
* sexually active
* identifies as male
* report HIV risk characterized by one or more of the following: 1) condomless anal or vaginal sex (receptive or penetrative) with a partner assigned male at birth (AMAB) of unknown HIV status in the last 6 months, 2) presence of rectal STI in the last 6 months, 3) condomless anal or vaginal sex with a known HIV-infected partner in the last 6 months (inclusive of partners who are undetectable), or 4) condomless anal or vaginal sex (receptive or penetrative) with casual partners assigned male at birth and endorsement of factors associated with not using PrEP based on my preliminary research with the MDPH (i.e., non-disclosure of same-sex behavior to provider, uninsured, history of incarceration, or lacking healthcare due to cost). For participants under the age of 18, condomless sex criteria can be met by having condomless oral sex.

Exclusion Criteria:

Those unable to complete consent in English and those with significant mental health diagnoses (e.g., uncontrolled psychosis) that would likely interfere with participation will be excluded and referred for treatment or alternative resources as necessary.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender or Transgender men or non-binary individuals assigned male at birth
Enrollment: 5 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
PrEP Use | 3 months
  Self-reported use of PrEP
PrEP Adherence | 6 months
  Dried blood spots

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No